CLINICAL TRIAL: NCT03812575
Title: The Use of Fractionated Exhaled Nitric Oxide in the Diagnosis and Assessment of Disease Activity of Eosinophilic Esophagitis
Brief Title: The Use of Fractionated Exhaled Nitric Oxide in the Diagnosis and Assessment of Disease Activity of Eosinophilic Esophagitis (Pilot)
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Tu Thanh Mai, Assistant Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-18-1019 (pilot)
Record Dates: First submitted 2019-01-18; First posted 2019-01-23 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Active eosinophilic esophagitis
- Eosinophilic esophagitis in remission
- No eosinophilic esophagitis

SUMMARY:
The purpose of the study is to evaluate of the relationships between fractionated exhaled nitric oxide, disease activity, and symptom severity in patients with eosinophilic esophagitis compared to those without eosinophilic esophagitis.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patient who will undergo esophagogastroduodenoscopy with biopsies at Children's Memorial Hermann Hospital, as part of the standard of care in the evaluation of EoE
* Able to perform the single-breath exhalation for the hand-held analyzer, NIOX MINO (Aerocrine, Sweden)
* Signed informed consent by a parent or legal guardian
* Signed assent form by the child/adolescent subjects 7-18 years of age

Exclusion Criteria:

* Past medical history of asthma, allergic rhinitis, IBD, parasitic infection, hay fever and any exposure to smoking (including secondhand smoke) because these disorders are known to affect the FeNO levels
* Active respiratory tract infections at the time of FeNO evaluation because this can affect the result of the FeNO as well
* Asthma questionnaire and/or Spirometry test consistent with asthma

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients will be recruited from the outpatient clinic of the Pediatric Gastroenterology Division of The University of Texas Health and Science Center at Houston.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Fractionated exhaled nitric oxide (FeNO) level | baseline (day of first endoscopy)
  The FeNO measurement will be performed using a hand-held analyzer, the NIOX MINO (Aerocrine, Sweden). During this non-invasive procedure the patient is asked to perform a 4-6 second single-breath exhalation into the NIOX MINO, which measures FeNO in 100s with an electrochemical sensor.
Fractionated exhaled nitric oxide (FeNO) level | at about 4-12 weeks (day of second endoscopy)
  The FeNO measurement will be performed using a hand-held analyzer, the NIOX MINO (Aerocrine, Sweden). During this non-invasive procedure the patient is asked to perform a 4-6 second single-breath exhalation into the NIOX MINO, which measures FeNO in 100s with an electrochemical sensor.

SECONDARY OUTCOMES:
Esophageal eosinophil counts as assessed by biopsy | baseline (day of first endoscopy)
Esophageal eosinophil counts as assessed by biopsy | at about 4-12 weeks (day of second endoscopy)
Serum eosinophil counts as assessed by complete blood count (CBC) | baseline (day of first endoscopy)
Disease-related symptoms severity as assessed by Pediatric Eosinophilic Esophagitis Symptom Severity (PEESS) version 2.0 questionnaire | baseline (day of first endoscopy)
  The range of total score is 0 to 100, with a higher score being indicative of more frequent and/or severe symptoms.
Disease-related symptoms severity as assessed by Pediatric Eosinophilic Esophagitis Symptom Severity (PEESS) version 2.0 questionnaire | at about 4-12 weeks (day of second endoscopy)
  The range of total score is 0 to 100, with a higher score being indicative of more frequent and/or severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Tu T Mai, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Josyabhatla R, Abrenica C, Mai T, Hashmi SS, Liu Y, Mosquera R, Van Arsdall M, Navarro F, Tchakarov A, Tatevian N, Wu G, Rhoads JM. Plasma Biomarkers and Fractional Exhaled Nitric Oxide in the Diagnosis of Eosinophilic Esophagitis. J Pediatr Gastroenterol Nutr. 2023 Jan 1;76(1):59-65. doi: 10.1097/MPG.0000000000003634. Epub 2022 Oct 11. PMID 36574003